CLINICAL TRIAL: NCT03158597
Title: Screening Pathogenic Genes Associated With Acute Myocardial Infarction and Studying Its Relevant Molecular Mechanism
Brief Title: Transcriptome Study of Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Responsible Party: Principal Investigator, Yan Li, Principal Investigator, Beijing Institute of Heart, Lung and Blood Vessel Diseases
Other Study IDs: 5172011
Record Dates: First submitted 2017-05-15; First posted 2017-05-18 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AMI
- Control

SUMMARY:
This study aims to compare whole-blood microarray gene-expression profiling between patients with acute myocardial infarction and normal participants without cardiovascular diseases. Firstly, screening differentially genes of mRNA to perform gene ontology and pathway analysis. Secondly, predicting target genes regulated by microRNA and constructing coexpression network with mRNA. Thirdly, biological function experiment of microRNA. Finally, revealing pathogenic mechanisms associated with acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* AMI patients:

  1. 20-50 years of age
  2. Symptoms of ischaemia
  3. New significant ST-segment-T wave changes in ECG and definitive diagnosis of non-ST elevation MI or ST elevation MI
  4. Cardiac troponin with at least one value above the 99th percentile upper reference limit
* Normal control participants:

  1. 20-50 years of age
  2. Normal ECG
  3. BMI <24kg/m2
  4. systolic blood pressure <140mmHg
  5. diastolic blood pressure <90mmHg
  6. Total cholesterol <200mg/dl (5.18mmol/L)
  7. Triglyceride <150mg/dl (1.70mmol/L)
  8. High density lipoprotein cholesterol >=40mg/dl (1.04mmol/L)
  9. Low density lipoprotein cholesterol <130mg/dl (3.37mmol/L)
  10. Fasting blood glucose <100mg/dl (5.6mmol/L)
  11. Not taking antihypertensive or hypolipidemic or hypoglycemic drugs

Exclusion Criteria:

1. Cardiac death with symptoms suggestive of myocardial ischaemia and presumed new ischaemic ECG changes, but death occurred before cardiac biomarkers were obtained, or before cardiac biomarker values would be increased
2. Prior myocardial infarction
3. Percutaneous coronary intervention related MI
4. Stent thrombosis associated with MI
5. Coronary artery bypass grafting related MI
6. Recurrent MI or reinfarction
7. Myocardial injury with necrosis caused by transcatheter aortic valve implantation or mitral clip or ablation of arrhythmias
8. Myocardial injury or infarction associated with heart failure
9. Myocardial infarction in the intensive care unit
10. Other diseases: previous history of ASCVD, cancer, rheumatoid arthritis, liver or kidney disease, myeloproliferative disorders, chronic inflammation, peripheral vascular disease
11. Not available informed consent

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: AMI patients will be selected from Emergency Department of Beijing An Zhen Hospital or Beijing Tong Ren Hospital.
  Normal control participants will be recruited from Health Examination Center of Beijing An Zhen Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of screening differentially expressed genes associated with acute myocardial infarction as measured by microarray | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Chaoyang, China